CLINICAL TRIAL: NCT05186402
Title: Predictive Factors of Morbidity and Mortality and Overall Survival of Patients With Gastric Cancer : a Case Series
Status: Completed | Type: Observational
Sponsor: Sylvestre KABURA (Other)
Responsible Party: Sponsor-Investigator, Sylvestre KABURA, Principal investigator, Centre Hospitalier Universitaire Ibn Rochd
Organization: Centre Hospitalier Universitaire Ibn Rochd (Other)
Other Study IDs: SKAHM2022
Record Dates: First submitted 2021-12-27; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Gastric Cancer; Mortality of Gastric Cancer; Overall Survival of Patients With Gastric Cancer
Keywords: gastric cancer mortality, gastric cancer treatment
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: Total or subtotal gastrectomy — Gastric resection with digestive continuity according Roux or Bilroth
  Other Names: Adjuvent chemotherapy

SUMMARY:
This is a retrospective study extending over a period of three years concerning patients with gastric adenocarcinoma hospitalized in the digestive cancer surgery and liver transplant service of the IBN ROCHD University Hospital Center in Casablanca. Evaluation from a series of 80 cases of gastric adenocarcinomas, follow-up to determine the prognostic factors influencing mortality, morbidity and survival.

ELIGIBILITY:
Inclusion Criteria:

* patients with gastric cancer

Exclusion Criteria:

* patients with benign tumors or other pathologies requiring gastric resection

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study enrolled all the patients who underwent gastric resection for gastric adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 30 months
  An overall survival of patients treated for gastric cancer

IPD SHARING:
Plan to Share IPD: Undecided